CLINICAL TRIAL: NCT05175963
Title: Surveillance Among Healthcare Workers for SARS-Coronavirus-2 Infection
Status: Completed | Type: Observational
Sponsor: Farzanah Laher (Other)
Responsible Party: Sponsor-Investigator, Farzanah Laher, Dr, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Other Study IDs: 200405
Record Dates: First submitted 2022-01-02; First posted 2022-01-04 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: COVID-19; SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- High Risk: Nurses (auxiliary nurses, enrolled nurses and professional nurses), medical doctors (interns, medical officers, registrars and consultants) and auxiliary/para-medical staff involved in the care of patients admitted for respiratory illnesses at Chris Hani Baragwanath Academic Hospital (CHBAH). This will include staff that have been assigned to work in:
  Internal Medicine: Staff working in the Ambulatory and Emergency Department, staff in the "pneumonia-admission" ward (ward 24), and staff in the COVID-19 confirmed case wards.
  Paediatrics: Staff involved in-hospital care of patients admitted to the dedicated "pneumonia ward" and COVID-19 cases wards.
  Intensive Care Unit: All medical staff working in the intensive care unit.
- Low Risk: Nursing and medical-doctor staff that are working in the neonatal high-care and intensive care unit; who are likely to be at lower risk from SARS-CoV-2 acquisition in the health-care facility compared to their peers listed in Group 1.
- Intermediate Risk: A third group, with a likely intermediate risk for hospital-facility based SARS-CoV-2 infection, are:
  VIDA staff involved in sample collection related to COVID-19, and laboratory personnel that will be involved in sample collection at VIDA.
  Nurses and medical doctors from the Obstetrics & Gynaecology.
- Mixed Risk: In 2021 with an eminent 3rd wave spreading across the country an additional group will be included comprising of any person working at CHBAH even if not in direct contact with patients.
- TND group: Any person working at CHBAH or Charlotte Maxeke Johannesburg Academic Hospital (CMJAH) and Helen Joseph Hospital (HJH) even if not in direct contact with patients.

SUMMARY:
This study aims to investigate the epidemiology of SARS-CoV-2 infection among: i) HCW who triage patients with suspected SARS-CoV-2 infection and provide care to COVID-19 patients; and ii) laboratory personnel who test clinical samples for SARS-CoV-2 infection. After the second wave of the pandemic enrolment will be widen to any person working at the study hospitals.

ELIGIBILITY:
Inclusion Criteria:

* HCWs of any staff category at the study hospitals.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any HCWs of any staff category at the study hospitals
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of symptomatic and asymptomatic SARS-CoV-2 infections among HCW. | 2020
  To determine the prevalence of symptomatic and asymptomatic PCR-confirmed SARS-CoV-2 infections among HCW using a systematic sampling strategy, coupled with investigation when clinically indicated.

SECONDARY OUTCOMES:
To define the duration of viral "shedding". | 2020
  To define the duration of "shedding" (using molecular based PCR methods) of SARS-CoV-2 in HCW who are identified to be infected with the virus.
To do sero-epidemiology assessment. | 2022
  To undertake serial sero-epidemiology studies on prevalence of SARS-CoV-2 antibodies among HCW.
To analyse immune responses to SARS-CoV-2 infection. | 2022
  To analyse immune responses (humoral and cell mediated) to SARS-CoV-2 infection.
To investigate the possibility of viral re-infection in this population during the study period. | 2022
  To investigate the possibility of viral re-infection during the different pandemic waves in this population during the study period.
To establish if common cold coronaviruses (CCCV) immunity confers protection against SARS-CoV-2 infection or disease severity | 2022
  To establish if common cold coronaviruses (CCCV) immunity confers protection against SARS-CoV-2 infection or disease severity by measuring antibodies to CCCV.
To evaluate COVID-19 vaccine effectiveness (VE) amongst HCWs, against any PCR-confirmed SARS-CoV-2 infection. | 2022
  To evaluate COVID-19 vaccine effectiveness (VE) amongst HCWs, against any PCR-confirmed SARS-CoV-2 infection.
To measure humoral and cell mediated immune responses to COVID-19 vaccines stratified by previous SARS-CoV-2 infection. | 2022
  To measure humoral and cell mediated immune responses to COVID-19 vaccines stratified by previous SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Chris Hani Baragwanath Academic Hospital, Johannesburg, GP, South Africa